CLINICAL TRIAL: NCT06437743
Title: Monitoring Nociception Using NoL Index and Its Implications in Reducing Opioid-Related Complications in Laparoscopic Abdominal Surgery
Brief Title: Monitoring Nociception Using NoL Index to Reduce Opioid-Related Complications in Laparoscopic Abdominal Surgery
Acronym: SIMONE
Status: Not yet recruiting | Type: Observational
Sponsor: Investigation Group Anesthesia, Resuscitation, And Perioperative Medicine of Aragon (Network)
Responsible Party: Sponsor
Other Study IDs: SIMONE001
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Opioid-related Complications
Keywords: Nociception, NoL Index, Opioids, Postoperative Complications, Laparoscopic Surgery
MeSH Terms: conditions — Postoperative Complications | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NoL Visible: Patients in this group will undergo laparoscopic abdominal surgery with the nociception level (NoL) monitor visible to the anesthesiologist. The NoL monitor provides an estimation of nociception through a multi-parameter sensor placed on the patient's finger. The anesthesiologist will adjust the doses of analgesic drugs based on the values observed on the NoL monitor, aiming to maintain the values between 10 and 25 during the surgery.
  Interventions: Device: Nociception Level (NoL) Monitor
- NoL Not Visible: Patients in this group will undergo laparoscopic abdominal surgery with the NoL monitor not visible to the anesthesiologist. The monitor will still be in place and collecting data, but its values will not be displayed during the surgery. The anesthesiologist will manage analgesia based on standard hemodynamic parameters such as heart rate and blood pressure, without access to the NoL values. The intervention includes the same standard anesthetic protocol as the NoL Visible group.
  Interventions: Device: Nociception Level (NoL) Monitor

INTERVENTIONS:
Device: Nociception Level (NoL) Monitor — The NoL Monitor (PMD-200) is a multi-parameter sensor device placed on the patient's finger to estimate nociception levels during surgery. It provides continuous, real-time feedback to the anesthesiologist on the patient's nociception, assisting in the optimization of analgesic drug administration. The monitor integrates parameters such as heart rate variability, skin conductance, and other physiological signals to compute the NoL index, which ranges from 0 to 100, with target values between 10 and 25 for optimal nociception management.
  Other Names: PMD-200

SUMMARY:
This study aims to determine if optimal intraoperative nociception monitoring using the NoL index can reduce postoperative complications related to opioid use in laparoscopic abdominal surgery. The hypothesis is that guided nociception monitoring decreases opioid-related complications and improves postoperative outcomes.

DETAILED DESCRIPTION:
The study is a prospective, observational cohort study conducted across multiple centers. It aims to evaluate the impact of intraoperative nociception monitoring on postoperative opioid-related complications. The study will involve two groups of patients undergoing laparoscopic abdominal surgery: one group with visible NoL monitoring and another with non-visible NoL monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for laparoscopic abdominal surgery
* Undergoing balanced general anesthesia
* ASA physical status I-III
* Signed informed consent

Exclusion Criteria:

* Refusal to participate
* Communication barriers
* Multimodal, opioid-free, or regional epidural anesthesia
* ASA IV or V
* Pregnant or breastfeeding women
* Open or emergency abdominal surgery
* Post-surgery transfer to ICU or Recovery Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients scheduled for elective laparoscopic abdominal surgery at participating hospitals. The population will consist of individuals who meet the inclusion criteria and have consented to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Postoperative Opioid-Related Complications | From the end of surgery up to 48 hours postoperatively
  The primary outcome measure will evaluate the incidence of postoperative opioid-related complications in patients undergoing laparoscopic abdominal surgery. Complications include nausea, vomiting, respiratory depression, and opioid-induced hyperalgesia. The study aims to determine if the use of the NoL monitor to guide intraoperative analgesia reduces these complications compared to standard hemodynamic monitoring.

SECONDARY OUTCOMES:
Intraoperative Opioid Consumption | During the surgical procedure
  This secondary outcome measure will assess the total amount of opioids administered during surgery. The comparison will be made between the group with visible NoL monitoring and the group with standard hemodynamic monitoring.
Postoperative Pain Scores | At 1, 6, 12, 24, and 48 hours postoperatively
  Postoperative pain levels will be measured using the Visual Analog Scale (VAS) at various time points post-surgery. The study will compare pain scores between the two groups to evaluate the effectiveness of NoL-guided analgesia.
Length of Hospital Stay | From admission to discharge, up to 7 days postoperatively
  This secondary outcome will measure the duration of hospital stay from admission to discharge following surgery. The aim is to determine if NoL-guided analgesia affects the length of hospitalization.

OTHER OUTCOMES:
Patient Satisfaction with Pain Management | At 48 hours postoperatively
  Patient satisfaction with pain management will be assessed using a standardized questionnaire. The goal is to compare satisfaction levels between the NoL visible group and the standard monitoring group.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Pascual-Bellosta, M.D, Ph.D, Prof., Principal Investigator — Miguel Servet University Hospital; Cristian Aragón-Benedí, M.D, Ph.D, Study Chair — Miguel Servet University Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers for this study.

REFERENCES:
- [Derived] Pascual-Bellosta AM, Aragon-Benedi C, Ortega-Lucea SM, Minguez-Braulio L, Buey-Aguilar M, Abad-Gurumeta A, Tamayo-Gomez E, Martinez-Ubieto J; SIMONE Trial Group. Monitoring of nociception by NoL Index and its implication in the reduction of opioid complications in laparoscopic abdominal surgery (SIMONE study): Protocol of a prospective, multicentre, observational cohort study. Rev Esp Anestesiol Reanim (Engl Ed). 2025 Jun;72(6):501729. doi: 10.1016/j.redare.2025.501729. Epub 2025 Feb 22. PMID 39993632